CLINICAL TRIAL: NCT07069335
Title: A Multi-centre, Open-Label, Randomized, Two-Stage, Two-treatment, Two-Period, Multiple-Dose, Crossover Bioequivalence Study to Evaluate the Pharmacokinetic Characteristics and the Safety Between Administration of BR2022 and BR2022-1 in Patients With Deleterious or Suspected Deleterious Germline BRCA-Mutated Advanced Ovarian Cancer
Brief Title: A Bioequivalence Study to Evaluate Pharmacokinetics and Safety of BR2022 and BR2022-1 in Patients With Deleterious or Suspected Deleterious Germline BRCA-Mutated Advanced Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-OLP-CT-101
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer
Keywords: BRCA-mutated; Ovarian Cancer; BR2022
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (TR) (Experimental): Subjects are randomized into two sequence groups (Sequence 1 and 2). In Sequence 1, subjects receive T (1d-7d) then R (8d-14d) T: Test treatment BR2022 (Olaparib 150.00mg) R: Reference treatment BR2022-1 (Olaparib 150 mg) Washout interval: None
  Interventions: Drug: Olaparib 150 MG
- Sequence 2 (RT) (Experimental): Subjects are randomized into two sequence groups (Sequence 1 and 2). In Sequence 2, subjects receive R (1d-7d) then T (8d-14d) T: Test treatment BR2022 (Olaparib 150.00mg) R: Reference treatment BR2022-1 (Olaparib 150 mg) Washout interval: None
  Interventions: Drug: Olaparib 150 MG

INTERVENTIONS:
Drug: Olaparib 150 MG — Subjects receive 600 mg per day, two tablets BID (total 4 tablets), oral administration
  Other Names: BR2022

SUMMARY:
This was a multicenter, open-label, randomized, crossover bioequivalence study to evaluate the pharmacokinetics and safety of BR2022 and BR2022-1 in Patients with deleterious or suspected deleterious germline BRCA-mutated advanced ovarian cancer.

DETAILED DESCRIPTION:
This study will be conducted in two stages. Stage 1 enrolls patients who have been taking BR2022-1 as existing therapy, and results will be evaluated before deciding whether to proceed with the Stage 2 part of the study and enroll more patients.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 19 -74 at the time of consent
2. Those who voluntarily signed the informed consent to participate in this study
3. Patients with deleterious or suspected deleterious germline or somatic BRCA-mutated advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer who have been taking stable doses of olaparib for more than 3 months before screening.

Exclusion Criteria:

1. Those who have a history of severe hypersensitivity to drugs that include the ingredients of the investigational product or have a history of clinically significant hypersensitivity reactions
2. Those who have gastrointestinal disorders (e.g., gastroesophageal reflux disease, gastrospasm, gastritis, gastrointestinal ulcers, Crohn's disease, etc.) or have had surgeries (excluding appendectomy or hernia surgery) that may affect the absorption of the investigational products
3. Those who are pregnant, suspected of pregnancy, or nursing

Ages: 19 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic variable - Cmax | From Day 6 to Day 7 after dose administration
  Maximum plasma concentration of BR2022 and BR2022-1
Pharmacokinetic variable - AUCtau | From Day 6 to Day 7 after dose administration
  Area under the drug concentration-time curve over the time interval from Day 6 to Day 7 after dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa District, South Korea

IPD SHARING:
Plan to Share IPD: No